CLINICAL TRIAL: NCT02596828
Title: Prospective Pilot Trial to Assess a Multimodal Molecular Targeted Therapy in Children, Adolescent and Young Adults With Relapsed or Refractory High-grade Pineoblastoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Regensburg (Other)
Responsible Party: Principal Investigator, Prof. Dr. med. Selim Corbacioglu, Professor Dr. med., University of Regensburg
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RIST-rPB-2015-P
Record Dates: First submitted 2015-10-28; First posted 2015-11-04 (Estimated); Last update posted 2021-08-05 (Actual); Status verified 2021-07

CONDITIONS: Pineoblastoma
Keywords: molecular targeted therapy; protein kinase inhibitor; mTOR Inhibitor; cytostatic topoisomerase-I-inhibitor; temozolomide; irinotecan; dasatinib; rapamycin
MeSH Terms: conditions — Pinealoma | interventions — Temozolomide; Irinotecan; Dasatinib; Sirolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- RIST (Experimental)
  Interventions: Drug: Temozolomide; Drug: Irinotecan; Drug: Dasatinib; Drug: Rapamycin

INTERVENTIONS:
Drug: Temozolomide — Pharmacotherapeutic Group: Antineoplastic agents - Other alkylating agents, ATC-Code: L01A X03 Excipients: Capsule content: Anhydrous lactose, Sodium starch glycolate Type A, Colloida anhydrous silica, Tartaric acid, Stearic acid. Capsule shell: Gelatine, Titanium dioxide (E171).
  Printing ink: Shellac Propylene glycol, Titanium dioxide (E171), Sunset yellow FCF Aluminium Lake (E110) Formulation: capsule, hard Route of Administration: orally; Temomedac hard capsules should be administered in the fasting state. The capsules must be swallowed whole with a glass of water and must not be opened or chewed
  Other Names: Temomedac
Drug: Irinotecan — Pharmacotherapeutic Group: cytostatic topoisomerase-I-inhibitor ATC-Code: L01XX19 Excipients: Sorbitol (E420), lactic acid, sodium hydroxid (to adjust the pH to 3.5), water for injection Formulation: concentrate for solution for infusion Route of Administration: intravenously
  Other Names: Irinomedac
Drug: Dasatinib — Pharmacotherapeutic Group: protein kinase inhibitor ATC-Code: L01XE06 Excipients: Tablet core: Lactose monohydrate, Cellulose, microcrystalline, Croscarmellose sodium, Hydroxypropyl cellulose, Magnesium stearate. Film-coating: Hypromellose, Titanium dioxide, Macrogol 400 Formulation: film coated tablet Route of Administration: orally. Patients should be instructed to swallow the tablets as a whole and not to split, chew, or crush them.
  Other Names: Sprycel
Drug: Rapamycin — Pharmacotherapeutic Group: Immunosuppressive agents - mTOR Inhibitors ATC-Code: L04A A10 Excipients: Polysorbat 80, Phosal 50 PG ((3-sn-Phosphatidyl)cholin from Soy beans, Propylenglycol, lipid acid mono- and -diglyzeride from Soy oil, Ethanol (1,5% bis 2,5%), Soy liid acid and Palmitoyl ascorbic acid) Formulation: Oral solution Route of Administration:orally
  Other Names: Rapamune

SUMMARY:
Children, adolescents and young adults with relapsed or treatment refractory pineoblastoma (rPB) represent a group of patients with dismal prognosis for whom a recommended standard salvage therapy is currently not available.

DETAILED DESCRIPTION:
The multimodal metronomic approach combining molecular targeted drugs (rapamycin and dasatinib) with conventional chemotherapy (irinotecan and temozolomide) will be investigated in a randomized fashion as new treatment strategy for patients with rPB. The intention is to assess the therapeutic benefit of molecular targeted drugs for the treatment of rPB.

The combination of irinotecan and temozolomide showed activity in the treatment of several solid organ tumors, brain tumors and neuroblastoma. In one study relapsed neuroblastoma (rNB) patients received a median of 5 courses of 5 days irinotecan and temozolomide every 3 to 4 weeks with a cumulative dose of 35% lower than in the RIST design. 33% had disease regression with 8% CR or PR. A phase II study in rNB also using irinotecan and temozolomide with a substantially lower intensity showed a response rate of 15%.

The combination of a mTOR inhibitor with a multi-kinase inhibitor demonstrated in preclinical studies a synergistic effect on cell cycle arrest, apoptosis and sensitization for radio- and chemotherapy. It is assumed that this combination of molecular targeted drugs with a tolerable conventional chemotherapy consisting of irinotecan and temozolomide can substantially improve the outcome of this patient population. A group of 20 rNB patients treated with the RIST therapy approach in a compassionate use setting showed an overall survival of 55% at a median of 80 weeks with a tolerable adverse event profile.

ELIGIBILITY:
Inclusion Criteria:

Patients with relapsed and refractory high-grade pineoblastome (=rPB) and all of the following criteria will be considered for admission to the clinical trial:

* Children, adolescents and young adults 0 months to 25 years
* Signed written informed consent (patient or his/her parents/legal guardian)
* Females of childbearing age must have a negative urine pregnancy test prior to starting the study drug. The first pregnancy test must be performed within 10-14 days prior to the start of the study drug and the second pregnancy test must be performed within 24 hours prior to the start of study drug. The subject may not receive the study drug until the investigator has verified that the results of these pregnancy tests are negative.
* Females of childbearing age must comply with the institutional standards of birth control with a pearl index <1%. Contraception must be started at least four weeks before the start of the investigational therapy.
* Females of childbearing age must be willing to abstain from breastfeeding for the duration of the clinical trial and for at least 30 days after discontinuation of the clinical trial.
* Males must agree not to father a child and must use latex condom during any sexual contact with women of childbearing age during and for 6 months after therapy ends or is stopped, even if they have undergone successful vasectomy.
* Willing and able to complete the clinical trial procedures, as described in the protocol
* Non-smoker for at least the previous 3 months. Smoking is not allowed during the entire study period
* Abstain from alcohol within the last 24 hours before screening and before admission to the clinical trial center as well as during the entire clinical trial. The regular daily ethanol intake has to be less than 20g/day for at least the previous three months.
* Patients are required to have an absolute neutrophil count (ANC) ≥500/µL, hemoglobin ≥8g/dL (transfusion permitted), and an unsupported platelet count ≥30,000/µL unless:

  * patient is refractory or relapsed early after primary therapy

Exclusion Criteria:

Patients presenting with any of the following criteria will not be included in this clinical trial:

* Pregnancy, nursing
* Patients who suffered from a thrombotic event and need anticoagulation (i.e. coumadine derivatives or low molecular weight heparin derivatives, LMWH)
* Patients with cardiac arrhythmias especially prolonged QT
* Patients with chronic inflammatory bowel diseases and/or bowel obstruction
* Patients with bilirubin serum levels 1,5 fold above the upper normal limit
* Vaccination with a live virus vaccine during the clinical trial
* Impaired liver function and/or impaired renal function (hepatic and renal index parameter two times above normal range; see below)
* Potentially unreliable subjects, probably non compliant subjects and those judged by the investigator to be unsuitable for the study
* Doubts about the patient's cooperation
* Any contraindications or known hypersensitivity to the IMPs or to any of the other components: (see SPC "Fachinformation")
* Known allergic reactions to the treatment medication
* Patients who were treated with radiation and/or chemotherapy for any other oncological condition
* Participation in any other interventional phase I to III trial
* Sexually active patients who refuse to use contraception according to the institutional requirements
* Patients with extremely poor general condition (Karnofsky or Lansky score <50%)
* Neutrophil count (ANC) <500/µL, hemoglobin <8g/dL (transfusion permitted), and an unsupported platelet count <30 000/µL
* 12-lead ECG with QTc>500 msec / QTc>60 msec baseline

  * Patients with hepatitis B reactivation

Ages: 0 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 4 (Actual)
Dates: Start 2016-04; Primary Completion 2021-04 (Actual); Study Completion 2021-04 (Actual)

PRIMARY OUTCOMES:
The primary endpoint is progression-free survival (PFS) | Time interval from date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 52 weeks
  According to:
  * Imaging criteria to
    * MRI, CT or
    * CSF evaluations or
  * date of death of any cause

SECONDARY OUTCOMES:
Overall survival (OS) | From the first course of the investigational treatment up to the end of the trial assessed to 52 weeks
  According to: questionnaire
Response to the investigational treatment after 4 and 8 courses of I/T and 1-year-follow-up in the RIST treatment arm | From the first course of the investigational treatment up to the end of the trial assessed to 52 weeks
  According to:
  • Imaging criteria to
  * MRI, CT or
  * CSF evaluations
Duration until adequate response to this treatment regimen | From the first course of the investigational treatment up to the end of the trial assessed to 52 weeks
  According to:
  • Imaging criteria to
  * MRI, CT or
  * CSF evaluations
Assessment of quality of life (Lansky and Karnofsky Scores) | From the first course of the investigational treatment up to the end of the trial assessed to 52 weeks
  According to:
  Lansky and Karnofsky Scores
Toxicity of this combination of drugs in children, adolescents and young adults with rNB - Assessment according to the latest version of the CTC criteria | From the first course of the investigational treatment up to the end of the trial assessed to 52 weeks
  Assessment according to the latest version of the CTC criteria. In particular due to the expected AE Profile:
  Myelosuppressive measures (RBC, PLT units) Infectious complications Gastrointestinal problems
Safety and tolerability of the investigational treatment - Assessment according to the latest version of the CTC criteria | From the first course of the investigational treatment up to the end of the trial assessed to 52 weeks
  Assessment according to the latest version of the CTC criteria. In particular due to the expected AE Profile:
  Myelosuppressive measures (RBC, PLT units) Infectious complications Gastrointestinal problems

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital of Regensburg, Regensburg, Germany